CLINICAL TRIAL: NCT02020291
Title: Phase I Dose Escalating Study to Evaluate the Safety, Tolerability, Anti-Tumour Activity and Pharmacokinetic and Pharmacodynamic Profiles of Foxy-5 in Patients With Metastatic Breast, Colon or Prostate Cancer
Brief Title: Phase I Study to Evaluate Safety, Tolerability, Anti-Tumour Activity and PK Profiles of Foxy-5 in Metastatic Breast, Colon or Prostate Cancer
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: WntResearch AB (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: SMR-2562
Record Dates: First submitted 2013-12-11; First posted 2013-12-24 (Estimated); Last update posted 2016-02-02 (Estimated); Status verified 2016-02

CONDITIONS: Metastatic Breast Cancer; Colorectal Cancer; Prostate Cancer
Keywords: Foxy-5; Wnt-5A
MeSH Terms: conditions — Breast Neoplasms; Colorectal Neoplasms; Prostatic Neoplasms | interventions — Foxy-5 peptide

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- Foxy-5 (Experimental): Slow infusion of lyophilised and reconstituted Foxy-5 three times weekly on Monday, Wednesday and Friday for three weeks.
  Interventions: Drug: Foxy-5

INTERVENTIONS:
Drug: Foxy-5

SUMMARY:
The Wnt proteins belong to a family of proteins that have been demonstrated to play a role in the formation and dissemination of tumours. The present project focuses on the critical role of the Wnt-5a protein in the pathobiological processes that lead to metastatic cancer disease.

WntResearch has identified a formylated 6 amino acid peptide fragment, named Foxy-5, which mimick the effects of Wnt-5a to impair migration of epithelial cancer cells and thereby acting anti-metastatic. The aim of the present clinical phase 1 trial is to establish the recommended dose for a clinical phase 2 study and thereby further develop Foxy-5 as a first in class anti-metastatic cancer drug. Foxy-5 is designed to inhibit the development of metastasis by reducing the motility of cancer cells and should thereby increase the survival rates of patients with solid malignant tumours.

ELIGIBILITY:
Inclusion Criteria:

* Males and females of at least 18 years of age
* Histologically/cytologically documented diagnosis of metastatic breast, colon or prostate cancer, refractory to standard therapy or for which no curative therapy exists
* Loss of or reduced Wnt-5a protein expression in primary or metastatic tumour cells, characterised by IHC analysis
* Eastern Cooperative Oncology Group (ECOG) performance status of <= 1
* Life expectancy of at least 3 months
* Unresectable disease, i.e. the metastases cannot be surgically removed with a curative intent
* >= 4 weeks must have elapsed since the patient has received any other IMP
* >=4 weeks must have elapsed since the patient has received any anti cancer treatment; including radiotherapy (except for single dose of palliative radiotherapy), cytotoxic chemotherapy, biologic agents or targeted therapy
* >= 2 weeks must have elapsed since any prior surgery or therapy with bone marrow stimulating factors
* Adequate haematological functions as defined by:
* Absolute neutrophil count >= 1.5 10E9/L
* Platelets >= 100 10E9/L
* Hemoglobin >= 5.6 mmol/L
* Adequate hepatic function as defined by:
* Total bilirubin <= 1.5 x the upper limit of normal (ULN)
* Aspartate aminotransferase (AST) <= 2.5 x ULN*
* Alanine aminotransferase (ALT) <= 2.5 x ULN*

  * For patients with liver metastasis adequate hepatic function is defined by AST <= 5 x ULN and ALT <= 5 ULN.
* Adequate renal function as defined by Serum creatinine <= 1,5 x ULN
* Provision of written informed consent
* Willingness and ability to comply with scheduled visits, treatment plans, laboratory tests and other study procedures
* Sexually active males and females of child-producing potential, must use adequate contraception (intrauterine devices, hormonal contraceptives (contraceptive pills, implants, transdermal patches, hormonal vaginal devices or injections with prolonged release) or diaphragm always with spermicidal jelly and a male condom) for the study duration and at least six months afterwards

Exclusion Criteria:

* Active uncontrolled bleeding or bleeding diathesis (e.g., active peptic ulcer disease)
* Any active infection requiring antibiotic treatment
* Known infection with human immunodeficiency virus (HIV) or hepatitis virus
* Active heart disease including myocardial infarction or congestive heart failure within the previous 6 months, symptomatic coronary artery disease, or symptomatic arrhythmias currently requiring medication
* Known or suspected active central nervous system (CNS) metastasis. (Patients stable 8 weeks after completion of treatment for CNS metastasis are eligible)
* Impending or symptomatic spinal cord compression or carcinomatous meningitis
* Requiring immediate palliative surgery and/or radiotherapy
* Pre-existing neuropathy, i.e., Grade >2 neuromotor or neurosensory toxicity
* Participation in other clinical studies within 4 weeks of first dose of study treatment
* History of severe allergic or hypersensitive reactions to excipients
* Pregnant or breastfeeding women
* Chronic immunosuppressant use (e.g. systemic steroids for treatment of autoimmune disease)
* History of second malignancy, including histologically confirmed diagnosis of malignant melanoma except for carcinoma in situ or basal cell carcinoma
* Severe or uncontrolled chronic or uncontrolled systemic disease (e. g. severe respiratory or cardiovascular disease)
* Other medications or conditions that in the Investigator's opinion would contraindicate study participation of safety reasons or interfere with the interpretation of study results

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 31 (Actual)
Dates: Start 2013-06; Primary Completion 2015-11 (Actual); Study Completion 2015-11 (Actual)

PRIMARY OUTCOMES:
Safety and tolerability of Foxy-5 | 1 year
  Assessment of adverse events and laboratory abnormalities

SECONDARY OUTCOMES:
Profile for the biomarker NGAL and the amount of circulating tumour cells before and after treatment with Foxy-5 | samples at pre-dose at day 1, pre-dose at day 12 and pre-dose at day 26
Profile for the biomarker 15-PGHD and the amount of circulating tumour cells before and after treatment with Foxy-5 | samples at pre-dose at day 1, pre-dose at day 12 and pre-dose at day 26
Maximum tolerated dose (MTD) | 1 year
  To determine the maximum tolerated dose (MTD) and dose-limiting toxicity (DLT) of Foxy-5.
  Assessment of adverse events and laboratory abnormalities
Area under the plasma concentration curve (AUC) of Foxy-5 | Plasma immediately prior to treatment, instantly after infusion, at 5, 15, 30, minutes 1, 3, 6, 8, 24, 48, 72 and 96 hours after infusion. In the Multiple dosing cycles on days 1+3+5 and 15+29
  The concentration of Foxy-5 in human biological samples will be measured with liquid chromatography with tandem mass spectrometry detection (LC-MS/MS).
Maximum observed plasma drug concentration (Cmax) of Foxy-5 | Plasma immediately prior to treatment, instantly after infusion, at 5, 15, 30, minutes 1, 3, 6, 8, 24, 48, 72 and 96 hours after infusion. In the Multiple dosing cycles on days 1+3+5 and 15+29
  The concentration of Foxy-5 in human biological samples will be measured with liquid chromatography with tandem mass spectrometry detection (LC-MS/MS).
Time to maximum observed plasma drug concentration (tmax) of Foxy-5 | Plasma immediately prior to treatment, instantly after infusion, at 5, 15, 30, minutes 1, 3, 6, 8, 24, 48, 72 and 96 hours after infusion. In the Multiple dosing cycles on days 1+3+5 and 15+29
  The concentration of Foxy-5 in human biological samples will be measured with liquid chromatography with tandem mass spectrometry detection (LC-MS/MS).
Terminal elimination half-life (t½) of Foxy-5 | Plasma immediately prior to treatment, instantly after infusion, at 5, 15, 30, minutes 1, 3, 6, 8, 24, 48, 72 and 96 hours after infusion. In the Multiple dosing cycles on days 1+3+5 and 15+29
  The concentration of Foxy-5 in human biological samples will be measured with liquid chromatography with tandem mass spectrometry detection (LC-MS/MS).
Total plasma clearance (CL) of Foxy-5 | Plasma immediately prior to treatment, instantly after infusion, at 5, 15, 30, minutes 1, 3, 6, 8, 24, 48, 72 and 96 hours after infusion. In the Multiple dosing cycles on days 1+3+5 and 15+29
  The concentration of Foxy-5 in human biological samples will be measured with liquid chromatography with tandem mass spectrometry detection (LC-MS/MS).
Volume of distribution (V) of Foxy-5 | Plasma immediately prior to treatment, instantly after infusion, at 5, 15, 30, minutes 1, 3, 6, 8, 24, 48, 72 and 96 hours after infusion
  The concentration of Foxy-5 in human biological samples will be measured with liquid chromatography with tandem mass spectrometry detection (LC-MS/MS).
Plasma concentration at steady state (Css) of Foxy-5 | Plasma immediately prior to treatment, instantly after infusion, at 5, 15, 30, minutes 1, 3, 6, 8, 24, 48, 72 and 96 hours after infusion. In the Multiple dosing cycles on days 1+3+5 and 15+29
  The concentration of Foxy-5 in human biological samples will be measured with liquid chromatography with tandem mass spectrometry detection (LC-MS/MS).
Drug accumulation ratio of Foxy-5 | Plasma immediately prior to treatment, instantly after infusion, at 5, 15, 30, minutes 1, 3, 6, 8, 24, 48, 72 and 96 hours after infusion
  The concentration of Foxy-5 in human biological samples will be measured with liquid chromatography with tandem mass spectrometry detection (LC-MS/MS).
mRNA expression and protein expression of Wnt-5a | Tumour biopsies obtained prior to day 1 and on day 12
Anti-tumour activity of Foxy-5 | Prior to Day 1 (-14 days is allowed) and at Day 12
  Voluntary tumour biopsies

CONTACTS AND LOCATIONS:
Locations (1):
- Oncology Department, Herlev Hospital, Herlev, Denmark